CLINICAL TRIAL: NCT06445868
Title: Construction and Preliminary Application of COM-B Based Sedentary Behavioural Booster Intervention Programme for Elderly Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Shuxian (Other)
Collaborators: Harbin Medical University (Other)
Responsible Party: Sponsor-Investigator, Liu Shuxian, researcher, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HMUDQ20231116221
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Knowledge (information support, changing health attitudes); Motivation (motivation to change sedentary behaviour and improve exercise compliance); Capacity (development of exercise plans to improve sedentary behaviour change); Opportunities (increasing the timing of exercise and creating opportunities for sedentary behaviour change); Behaviour (monitoring and reinforcing sedentary behaviour change)
  Interventions: Other: Sedentary behaviour intervention
- control group (No Intervention): Routine nursing education

INTERVENTIONS:
Other: Sedentary behaviour intervention — COM-B-based development of specific sedentary behavioral interventions to reduce sedentary time, promote healthy activity, and improve quality of life in older stroke patients
  Arms: intervention group

SUMMARY:
Explore the application effect of the sedentary behaviour intervention program for elderly stroke patients based on the COM-B model.

DETAILED DESCRIPTION:
The goal of this clinical trial is to text about in the application effect of the sedentary behaviour intervention program for elderly stroke patients based on the COM-B model. The main question it aims to answer are:

* Changes in sedentary behaviour in elderly stroke patients Participants will received a 12-week sedentary behaviour intervention programme.

Researchers will compare differences in sedentary behaviour between routine care control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for cerebral infarction and cerebral hemorrhage in the Diagnostic Points for Various Major Cerebrovascular Diseases in China 2019 issued by the Cerebrovascular Disease Group of the Neurology Branch of the Chinese Medical Association;
* Age ≥60 years;
* National Institute of Health stroke scale (NIHSS) score <5 (i.e., mild stroke), stable vital signs, and able to cooperate with the survey;
* Total sedentary time ≥6 hours/day measured using the International Physical Activity Questionnaire;
* Resident for ≥6 months in the community residents;
* Patients or under the guidance of others can use WeChat.

Exclusion Criteria:

* Functional ambulation category scale (FAC) score <2;
* serious myocardial infarction, cerebral hemorrhage and pulmonary embolism in the acute stage of the need to limit the activities of the situation;
* is participating in other physical activity or sedentary behavioral intervention programs;
* severe muscle weakness, fractures and other diseases resulting in limited physical activity;
* serious mental disorders such as schizophrenia or dementia resulting in severe cognitive impairment;
* speech and communication disorders.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
sedentary time | baseline (T0), 12-week post-intervention (T1), and 8-week follow-up (T2).
  International Physical Activity Questionnaire (IPAQ) Sedentary behavior and physical activity levels were assessed using the International Physical Activity Questionnaire (IPAQ), which was developed by the International Physical Activity Measurement Working Group (IPAMWG) in 2001, with the coefficients for sedentary behavior and validity scale correlation coefficients of 0.887 and 0.760 for sedentary behavior and 0.779 and 0.718 for physical activity, respectively. In this questionnaire, the metabolic equivalent of walking was 3.3, moderate activity intensity was 4.0, and high intensity activity was 8.0. The formula for calculating sedentary time was: sedentary time per day = (weekday sitting time x 5 + weekend sitting time x 2)/7
Social Support | baseline (T0), 12-week post-intervention (T1), and 8-week follow-up (T2).
  Social Support Rating Scale (SSRS) This scale is mainly used for the evaluation of individual social support status, with 10 entries, including 3 dimensions of subjective support, objective support and utilization of support. The scoring method is the sum of the scores of each entry, and the higher the score, the higher the level of social support. The scale reliability coefficient was 0.896.
Depression | baseline (T0), 12-week post-intervention (T1), and 8-week follow-up (T2).
  The Self-Rating Depression Scale (SDS) Self-Rating Depression Scale (SDS) is a 20-item self-rating scale, with scores of 1, 2, 3, and 4 for each item, and the sum of the scores of all items ranging from 53-62 indicating mild depression; 63-72 indicating moderate depression; and more than 72 indicating severe depression. The higher the total score, the more severe the depression. The Cronbach's alpha coefficient of the scale was 0.920.
Exercise Adherence | baseline (T0), 12-week post-intervention (T1), and 8-week follow-up (T2).
  Functional Exercise Adherence Scale for Stroke Patients (Questionnaire of Exercise Adherence, EAQ) The EAQ was developed by Beilei Lin in 2013 to assess patients' adherence to rehabilitation exercises. It contains 14 entries divided into 3 dimensions (physical participation in exercise, exercise effect monitoring and active seeking of exercise advice adherence), with each entry scored on a scale of 1 to 4. The total score of the scale ranges from 14 to 56, and the adherence index is the percentage value of the patient's measured score to the maximum score of the scale (56). The level of patient adherence was judged according to the adherence index: ≤50% = low level, 50% to 75% = medium level, and ≥75% = high level. The scale had good content validity (0.95), structural validity and validity scale validity, and high retest reliability (ICC: 0.778-0.850) and internal consistency (Cronbach's alpha coefficient: 0.923).
Ability to perform activities of daily living | baseline (T0), 12-week post-intervention (T1), and 8-week follow-up (T2).
  Modified Barthel Index Scale (MBI) The MBI scale was made in 1989 by Canadian scholars Shah and Vanchay, who subdivided the BI scale into 5 levels.The MBI scale[117] contains 10 basic activities of daily living (ADLs) such as dressing, grooming, eating, bathing, walking, transferring from bed and chair to toilet, etc., and is divided into 5 levels according to the degree of independence from 1-5, with the lowest being 1 and the highest being 5, which is determined and scored out of 100 points according to the completion of the patient's performance. The higher the score, the better the ability to perform activities of daily living.
10 meter maximum walking speed | baseline (T0), 12-week post-intervention (T1), and 8-week follow-up (T2).
  10 meter maximum walking speed (10 mMWS) The 10m maximum walking speed can reflect the patient's walking speed and walking functional status. First, a 16-meter straight line is drawn on a smooth surface, with markings at 3 and 13 meters. Let the patient walk along this straight line, assistive devices can be used, the timing starts when they reach 3 meters and ends at 13 meters, the time needed is recorded and the step speed is calculated at the same time, in this study, the test was done 3 times and the average value was taken, the faster the speed represents the better the walking ability and the slower the worse.